CLINICAL TRIAL: NCT02071004
Title: A PHASE 1, OPEN LABEL, SINGLE DOSE STUDY, TO ASSESS THE SAFETY AND TOLERABILITY OF A SINGLE IV DOSE OF DS-1040B AFTER 5 DAYS OF ASPIRIN TREATMENT IN HEALTHY SUBJECTS
Brief Title: DS1040b/Aspirin Drug/Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DS1040-A-E102
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2014-02

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Other): Dispersible tablet, 300mg & 75 mg, once daily for 5 days
  Interventions: Drug: Aspirin
- DS-1040b (Experimental): IV of 6 mg given once over 30 minutes
  Interventions: Drug: DS-1040b

INTERVENTIONS:
Drug: DS-1040b — IV of 6 mg given once over 30 minutes
  Arms: DS-1040b
Drug: Aspirin — Dispersible tablet, 300mg & 75 mg, once daily for 5 days
  Arms: Aspirin

SUMMARY:
This is a phase 1, open label, single dose study, after 5 days of aspirin treatment, in healthy male and female subjects. It is hypothesized that co-administering DS-1040b with aspirin at steady state will be safe and well tolerated by healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, aged 18 to 45 years.
* A body mass index (BMI, or Quetlet index) in the range of 18.0 to 30.0 kg/m2, and weighing between 50 and 100 kg at screening.
* Male subjects have to agree to contraception (condom with spermicide) in addition to having their female partner (if of child-bearing potential) use another form of contraception (e.g., an intrauterine device, diaphragm with spermicide, oral contraceptive, injectable, or sub dermal hormonal implant) from the first dose until 16 weeks following the last dose administration. Also, the male subjects must not donate sperm after the study for a period of four months.
* All women must have a negative serum pregnancy test at screening and a negative urine pregnancy test at admission (Day -1). Women must be of non-childbearing potential either: Surgically sterile (i.e., bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing) or naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing, with a follicle stimulating hormone (FSH) level at screening of ≥ 40 mIU/mL.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the ICF, and after having the opportunity to discuss the trial with the Investigator or his delegate.
* Willingness to give written consent to have data entered into The Overvolunteering Prevention Scheme.
* Willing to abstain from grapefruit/grapefruit juice and Seville oranges from 7 days before the first dose and throughout the study.
* Willing to refrain from consuming food or beverages containing caffeine/xanthine starting 24 hours prior to check-in on Day -1.

Exclusion Criteria:

* Clinically relevant abnormal history, including cardiovascular, haematologic, pulmonary, hepatic, renal, gastrointestinal, connective tissue disease, uncontrolled endocrine/metabolic, oncologic (within the last 5 years), neurologic (including previous transient ischemic attack or stroke), and psychiatric diseases, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* History of a serious reaction to any medicine.
* History of major bleeding, stomach ulcer, Raynaud's disease, major trauma, or major surgical procedure of any type within 6 months of dosing.
* History of minor bleeding episodes such as epistaxis, rectal bleeding (spots of blood on toilet paper), and gingival bleeding within 3 months before the study treatment.
* Familial or documented or suspected coagulopathy and haemoglobinopathy.
* Females with a history of dysfunctional uterine bleeding, including history of menorrhagia, metrorrhagia, or polymenorrhea.
* History of an operation (e.g. stomach bypass), or a condition that could affect how the body handles or absorbs medicines.
* History of gastro-oesophageal reflux disease.
* Females who are breastfeeding.
* Positive urine or faecal occult blood test at screening or admission (Day -1 or day 1).
* Bleeding time > 9.5 minutes at screening).
* aPTT, PT, INR, or platelet count outside the limit of normal of the clinical laboratory's reference range at screening.
* Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 (based on Modification of Diet in Renal Disease [MDRD] equation).
* Positive test for hepatitis B, hepatitis C, HIV1 & HIV2.
* QTcF interval duration > 430 msec for males and 450 msec for females, obtained as an average from the 3 ECG measurements on the triplicate screening ECGs.
* Abnormal waveform morphology on any of the ECGs at screening at admission that would preclude accurate measurement of the QT interval duration.
* Physical trauma, dental extraction, surgery, or a significant illness within 4 weeks before the first dose.
* History or presence of keloid, hyperpigmentation, or other adverse reaction to skin injury or surgery.
* Use of any prescribed or non-prescribed (over-the-counter [OTC]) systemic medications (including anticoagulants or antiplatelet medications), topical medications, or herbal supplements within 14 days before the first dose (excluding paracetamol ≤ 2 g/day). St. John's Wort (hypericin) must not have been taken for at least 30 days before the first dose.
* Donated or lost > 400 mL of blood or plasma during 3 months before the first dose on Day 1.
* Donation of blood, plasma, platelets, or any other blood components during the 3 months before the trial, or unwilling to abstain from doing so during the study and for 3 months after receipt of trial medication.
* Participated in a clinical study involving administration of an investigational drug, or a marketed drug within 90 days before administration of the first dose.
* Male subjects who consume more than 21 units of alcohol per week or female subjects who consume more than 14 units of alcohol per week (1 unit of alcohol equals 1/2 pint of beer, a glass of wine, or 1 measure of spirits) or those subjects who have a significant history of alcoholism or drug/chemical abuse within the last 2 years.
* Use of tobacco products or nicotine-containing products within 3 months before the first dose.
* Positive results on tests for drugs of abuse, carbon monoxide, or alcohol at screening or admission.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by General Practitioner (GP) to volunteer entering the trial.
* Known aspirin allergy or intolerance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
bleeding time | day 0 to day 5 after dosing
  To assess the safety (including bleeding time) and tolerability of a single IV dose of DS-1040b following 5 days aspirin treatment in healthy subjects

SECONDARY OUTCOMES:
change in D-dimer level | day 0 - day 5 after dosing
  To assess the effect of a single IV dose of DS-1040b following 5 days aspirin treatment on D-dimer levels
Cmax | Days 5, 6, and 7 after dosing
  Plasma concentration time data of DS-1040a (the free form of DS-1040b) will be analyzed using non-compartmental methods. The following parameters will be estimated and reported:
  .
Tmax | Days 5, 6, and 7 after dosing
  Plasma concentration time data of DS-1040a (the free form of DS-1040b) will be analyzed using non-compartmental methods. The following parameters will be estimated and reported:
AUC | Days 5, 6, and 7 after dosing
  Plasma concentration time data of DS-1040a (the free form of DS-1040b) will be analyzed using non-compartmental methods. The following parameters will be estimated and reported:
half-life | Days 5, 6, and 7 after dosing
  Plasma concentration time data of DS-1040a (the free form of DS-1040b) will be analyzed using non-compartmental methods. The following parameters will be estimated and reported:

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Limsakun T, Dishy V, Mendell J, Pizzagalli F, Pav J, Kochan J, Vandell AG, Rambaran C, Kobayashi F, Orihashi Y, Warren V, McPhillips P, Zhou J. Safety and Pharmacokinetics of DS-1040 Drug-Drug Interactions With Aspirin, Clopidogrel, and Enoxaparin. J Clin Pharmacol. 2020 Jun;60(6):691-701. doi: 10.1002/jcph.1568. Epub 2020 Feb 27. PMID 32106339